CLINICAL TRIAL: NCT03406949
Title: A Phase 1, Open Label, Dose Escalation Study of MGD009, a Humanized B7-H3 x CD3 DART® Protein, in Combination With MGA012, an Anti-PD-1 Antibody, in Patients With Relapsed or Refractory B7-H3-Expressing Tumors
Brief Title: MGD009/MGA012 Combination in Relapsed/Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD009-02
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: 3+3+3 dose escalation design followed by Cohort Expansion Phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- obrindatamab + retifanlimab (Experimental): B7-H3 x CD3 DART protein + anti-PD-1 antibody
  Interventions: Biological: obrindatamab; Biological: retifanlimab

INTERVENTIONS:
Biological: obrindatamab — B7-H3 x CD3 DART protein
  Other Names: MGD009
Biological: retifanlimab — anti-PD-1 antibody
  Other Names: INCMGA00012; MGA012

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics (PK) pharmacodynamics and preliminary antitumor activity of obrindatamab administered in combination with retifanlimab in patients with B7-H3- expressing tumors.

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, dose escalation, and cohort expansion study designed to characterize the safety, tolerability, PK, pharmacodynamics, immunogenicity, and preliminary antitumor activity of the combination of obrindatamab and retifanlimab, each of which is administered by IV infusion. The study consists of a Dose Escalation Phase to determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) (if no MTD is defined) of the combination, followed by a Cohort Expansion Phase to further define the safety and initial antitumor activity of the combination with the doses established in the Dose Escalation Phase. Patients with B7-H3-expressing unresectable, locally advanced, or metastatic solid tumors of any histology will be enrolled in the Dose Escalation Phase. Following the establishment of an MTD, additional patients with specific tumor types will enroll in the Cohort Expansion Phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven, unresectable locally advanced or metastatic solid tumors of any histology that test positive for B7-H3 expression on tumor cells or vasculature for whom no approved therapy with demonstrated clinical benefit is available. For all tumor types, the requirement for previous systemic therapy may be waived if a patient was intolerant of or refused standard first-line therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Measurable disease, with the exception of prostate cancer
* Tissue specimen available for B7-H3 and PD-L1 expression testing
* Acceptable laboratory parameters
* Patients who have previously received an immune checkpoint inhibitor (e.g., anti- PD-L1, anti-PD-1, anti-CTLA-4) prior to enrollment must have toxicities related to the checkpoint inhibitor resolved to ≤ Grade 1 or baseline (prior to the checkpoint inhibitor) to be eligible for enrollment. Patients who experienced previous hypothyroidism toxicity on a checkpoint inhibitor are eligible to enter study regardless of Grade resolution as long as the patient is well controlled on thyroid replacement hormones.

Exclusion Criteria:

* Patients with history of prior central nervous system (CNS) metastasis must have been treated, must be asymptomatic, and must not have any of the following at the time of enrollment:

  1. No concurrent treatment for the CNS disease (e.g. surgery, radiation, corticosteroids >10 mg prednisone/day or equivalent)
  2. No progression of CNS metastases on MRI or CT for at least 14 days after last day of prior therapy for the CNS metastases
  3. No concurrent leptomeningeal disease or cord compression
* Patients with any history of known or suspected autoimmune disease with the specific exceptions of vitiligo, resolved childhood atopic dermatitis, psoriasis not requiring systemic treatment (within the past 2 years), and patients with a history of Grave's disease that are now euthyroid clinically and by laboratory testing
* Treatment with any, investigational therapy within the 4 weeks prior to the initiation of study drug administration
* Treatment with any systemic chemotherapy within 3 weeks
* Treatment with radiation therapy within 2 weeks
* History of allogeneic bone marrow, stem-cell, or solid organ transplant
* Treatment with systemic corticosteroids (> 10 mg per day prednisone or equivalent) or other immune suppressive drugs within 2 weeks
* Clinically significant cardiovascular or pulmonary disease
* Evidence of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study drug. Patients requiring any systemic antiviral, antifungal, or antibacterial therapy for active infection must have completed treatment no less than one week prior to the initiation of study drug.
* Known history of positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome
* Known history of hepatitis B or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.03 | 30 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit.
MTD/MAD | 18 months
  Maximum Tolerated or Administrated Dose of obrindatamab and retifanlimab

SECONDARY OUTCOMES:
AUC | 30 months
  Area Under the Plasma Concentration versus Time Curve of obrindatamab and retifanlimab
Cmax | 30 months
  Maximum Plasma Concentration of obrindatamab and retifanlimab
Tmax | 30 months
  Time to reach maximum (peak) plasma concentration of obrindatamab and retifanlimab
Ctrough | 30 months
  Trough plasma concentration of obrindatamab and retifanlimab
CL | 30 months
  Total body clearance of the drug from plasma of obrindatamab and retifanlimab
Vss | 30 months
  Apparent volume of distribution at steady state of obrindatamab and retifanlimab
t1/2 | 30 months
  Terminal half life of obrindatamab and retifanlimab
ADA | 30 months
  Percent of patients with anti-drug antibody to obrindatamab and retifanlimab
Anti-tumor activity | 30 months
  Conventional Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-related response criteria (irRECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Eck, M.D., Study Director — MacroGenics
Locations (10):
- United States (10):
  - City of Hope Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START (South Texas Accelerated Research Therapeutics) - Midwest, Grand Rapids, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia